CLINICAL TRIAL: NCT02617030
Title: Developing a Program for Transition to Adult Care for Youth With Chronic Conditions : a Mixed Method Study
Acronym: TRANSAD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS 2013-NI 14003
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2018-02

CONDITIONS: Transition Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigation in 3 steps the transition of young people with chronic diseases. FIRST STEP: qualitative survey. Interviews with carers, young people and parents. Chronic Diseases studied: epilepsy, HIV, sickle cell disease, obesity. SECOND STEP: Delphi consensus survey. Vote on internet : carers, patients' associations, young people and family. Chronic Diseases studied: all. THIRD STEP: validation survey. Vote on internet : young people. Chronic Diseases studied: all.

ELIGIBILITY:
Inclusion Criteria:

* Youth with chronic diseases after transfer to adult care
* Parents or guardians of these youth.
* Professionals caregivers from pediatric services and adult services involved in transition

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Youth with chronic diseases after transfer to adult care
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Agreement rate for each component of the transition program defined | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gottot, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France

REFERENCES:
- [Background] Le Roux E, Mellerio H, Guilmin-Crepon S, Gottot S, Jacquin P, Boulkedid R, Alberti C. Methodology used in comparative studies assessing programmes of transition from paediatrics to adult care programmes: a systematic review. BMJ Open. 2017 Jan 27;7(1):e012338. doi: 10.1136/bmjopen-2016-012338. PMID 28131998
- [Result] Le Roux E, Gottot S, Aupiais C, Girard T, Teixeira M, Alberti C. Professional's Perspectives on Care Management of Young People with Perinatally Acquired HIV during Transition: A Qualitative Study in Adult Care Setting. PLoS One. 2017 Jan 23;12(1):e0169782. doi: 10.1371/journal.pone.0169782. eCollection 2017. PMID 28114376
- [Result] Le Roux E, Mellerio H, Jacquin P, Bourmaud A, Guilmin-Crepon S, Faye A, Matheron S, Boulkedid R, Alberti C. Practical generic guidelines for paediatric-to-adult transition for adolescents with chronic disease. Eur J Public Health. 2019 Jun 1;29(3):442-448. doi: 10.1093/eurpub/cky258. PMID 30535247